CLINICAL TRIAL: NCT02734576
Title: Venous Sinus Stenting To Treat Intractable Pulsatile Tinnitus Caused By Venous Sinus Stenosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to positive interim results.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1508016520
Record Dates: First submitted 2016-03-30; First posted 2016-04-12 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Tinnitus; Pulsatile Tinnitus; Venous Sinus Stenosis; Dural Sinus Stenosis
Keywords: Venous Sinus Stenting; Dural Sinus Stenting
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Venous Sinus Stenting (Experimental): Venous sinus stenting is the experimental procedure being tested in this protocol and consists of placing a stent into the narrowed veins of the brain. Under general anesthesia, a catheter will be inserted through a vein the upper part of the leg (groin area) and guided through the veins all the way to neck and the head. Then, a balloon will be advanced through the catheter and positioned across the stenosis. The balloon will be carefully inflated for a few seconds. This process is called angioplasty and will partially re-open the narrowing, making placement of the stent easier. The balloon will be removed and then the stent will be advanced through the catheter in neck across the stenosis and carefully deployed. After the procedure, the participants will stay in the intensive care unit for 24 hours for observation
  Interventions: Device: Venous Sinus Stenting with the Precise Pro Stent

INTERVENTIONS:
Device: Venous Sinus Stenting with the Precise Pro Stent — Enrolled patients will undergo a minimally invasive procedure that involves placement of a stent in the cerebral venous sinuses (large veins of the brain).

SUMMARY:
There have been few published studies that examine the efficacy and safety of endovascular treatments on patients with pulsatile tinnitus with venous stenosis. Despite the limited experience with venous sinus stenting to treat pulsatile tinnitus, preliminary results show that venous sinus stenting could represent a viable alternative for refractory pulsatile tinnitus patients with venous sinus stenosis. The purpose of this study is to evaluate the safety and efficacy of this procedure in a controlled fashion, using strict inclusion and exclusion criteria, and long-term clinical and imaging follow-up. The investigators hope to provide robust data regarding the safety and efficacy of venous sinus stenting for patients with pulsatile tinnitus.

DETAILED DESCRIPTION:
WHAT IS INVOLVED IN THE STUDY?

A. Screening process - not experimental:

Patients with pulsatile tinnitus, evidence of narrowing of the large veins of the brain, and failure of prior conservative treatment will be considered for enrollment. All patients will undergo the standard of care evaluation for tinnitus by a specialist physician for diseases of the ear (Ear, Nose and Throat [ENT] physician or otorhinolaryngologist). If it is determined that the narrowing of the large veins of the brain ("dural venous sinuses") is the most likely etiology for the tinnitus, then the possibility of enrollment in the trial will be discussed. Imaging studies of the head and temporal bone will be performed in order to further confirm venous sinus stenosis as the etiology of the pulsatile tinnitus and to rule out other possible causes. Additionally, patients will answer the questions listed on the Tinnitus Handicap Inventory questionnaire.

During the screening process, investigators will review the results of tests that are not experimental and are performed as part of participants' routine care. In other words, these tests are performed regardless of participation in the study and are termed "standard procedures".

B. Participating in the study:

Participating in the trial means that the participants will undergo an experimental procedure called "venous sinus stenting" to open up the narrowing in the vein that is causing the tinnitus. This procedure requires taking two blood thinners called aspirin and Plavix. Both blood thinners will be initiated 1 week prior to the procedure and continued for 1 month after the procedure. At that time the Plavix will be stopped and aspirin will be continued for 11 more months (total of 12 months).

- Direct Retrograde Cerebral Venography (DRCV) and Manometry: A DRCV is a non-experimental procedure to look at the veins of the brain. This procedure is done by inserting a catheter (soft plastic tube) through a vein in the groin (upper leg) and guide it though the veins all the way to the neck. It is done under local anesthetic and moderate sedation. After placing the catheter in the neck, a special dye (contrast) is injected through this catheter into the veins, while X-ray cameras take multiple pictures of the veins. Then, a smaller catheter is further advanced to the area of narrowing and by this catheter investigators will measure the blood pressure at that point. This helps us to identify the severity of the narrowing. If the pressure before and after the narrowing is significantly different, then the investigators will continue with the placement of the stent in order to reopen the narrowing.

- Venous Sinus Stenting (experimental): Venous sinus stenting is the experimental procedure being tested in this protocol and consists of placing a stent into the narrowed veins of the brain. The participants will be placed under general anesthesia because it is important to not move at all during the procedure. A catheter will be inserted through the upper part of the leg (groin area) and guided through the veins all the way to neck. Then, a balloon will be advanced through the catheter and positioned across the stenosis. The balloon will be carefully inflated for a few seconds. This process is called angioplasty and will partially re-open the narrowing, making placement of the stent easier. The balloon will be removed and then the stent will be advanced through the catheter in neck across the stenosis and carefully deployed.

- Post-procedure Care: After the procedure, participants will stay in the intensive care unit for 24 hours for observation.

C. Follow-up period:

There will be no experimental procedure or test during the follow-up period. The following office visits and standard tests will be performed to evaluate the effects of the study intervention.

- Office visits: Office visits and neurological evaluation will be performed at 1, 6, 12, and 24 months after study intervention. At this time, participants will also fill the Tinnitus Handicap Inventory Questionnaire. The visits will be about 45 min.

- Audiometric assessment: An audiometric assessment will be performed at 3 months after the stenting procedure in order to assess inner ear function.

- Non-invasive imaging studies: Magnetic Resonance Venogram (MRV) is a special Magnetic Resonance Imaging (MRI) scan with injection of a dye through a vein in the arm that will allow investigators to check whether the stent is still open without new narrowing. It will be performed 12 months after the venous sinus stenting procedure. If there is clinical concern about stent patency, an expedited or intermediate MRV will be performed. If MRV is contraindicated, Computed Tomographic Venogram (CTV) will be performed instead.

D. Medications:

For the purpose of the study, the participants need to take antiplatelet drugs ("blood thinners") that are necessary to prevent formation of clot in the stent. This is a standard precaution for every stent procedure. The participants will take two drugs (called aspirin and Plavix) for 1 month and then aspirin alone for 11 more months (total time on aspirin is 12 months). It is essential that the drugs are taken every day as prescribed. As these drugs are dangerous during pregnancy, if the participant is a woman of childbearing age, then should discuss this issue with her physician, and avoid becoming pregnant during the 12 months that these drugs are needed.

ELIGIBILITY:
Inclusion Criteria:

* Severe or catastrophic venous pulsatile tinnitus defined as Grades 4 or 5 on Tinnitus Handicap Inventory
* 50% or more stenosis of the lateral venous sinus on Magnetic Resonance Venogram (MRV) or Computed Tomographic Venogram (CTV_, ipsilateral to the side of more severe tinnitus
* Failure of conservative or non-surgical therapies (including sound therapy, sound masking, hearing aids, tinnitus retraining (desensitization) therapy. Failure is defined as Grades 4 or 5 on the Tinnitus Handicap Inventory despite prior treatments that have lasted for at least 3 months.

Exclusion Criteria:

* Non-pulsatile tinnitus
* Contra-indication to iodinated contrast
* Contra-indication to antiplatelet therapy
* Contra-indication to general anesthesia
* Pregnancy or plans for immediate pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athos Patsalides, MD MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital/ Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Venous Sinus Stenting: Venous sinus stenting is the experimental procedure being tested in this protocol and consists of placing a stent into the narrowed veins of the brain.
Period: Overall Study
Arm/Group | Venous Sinus Stenting
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Venous Sinus Stenting
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete or Near-complete Resolution of Tinnitus
Description: Tinnitus will be measured by: No, slight, mild, or moderate (Grades 1, 2, and 3) on Tinnitus Handicap Inventory.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Sinus Stenting
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Change in Number of Patients With Improvement of More Than One Grade in the Tinnitus Handicap Inventory Questionnaire
Description: Tinnitus will be measured by: No, slight, mild, or moderate (Grades 1, 2, and 3) on Tinnitus Handicap Inventory.
Time Frame: 1, 6, 12, and 24 months after stent placement.
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Sinus Stenting
Number analyzed (Participants) | 10
Participants | 10

3. Secondary Outcome: Number of Subjects With Clinical Recurrence of Their Tinnitus
Description: Clinical recurrence is if "No" tinnitus has changed back to "Slight, Mild or "Moderate."
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Sinus Stenting
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Number of Subjects With Long-term Patency of the Stent
Description: A subject is considered to have long-term patency if there is 100% patency of the stent at 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Sinus Stenting
Number analyzed (Participants) | 10
Participants | 10

5. Secondary Outcome: Number of Adverse Events Probably or Possibly Related to the Treatment
Time Frame: 24 months
Measure: Number; unit: adverse events
Arm/Group | Venous Sinus Stenting
Number analyzed (Participants) | 10
adverse events | 0

6. Secondary Outcome: Number of Severe Adverse Events Probably or Possibly Related to the Treatment
Time Frame: 24 months
Measure: Number; unit: severe adverse events
Arm/Group | Venous Sinus Stenting
Number analyzed (Participants) | 10
severe adverse events | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Any cause of disability.
Arm/Group | Venous Sinus Stenting
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT02734576/Prot_001.pdf